CLINICAL TRIAL: NCT01792479
Title: An Open Label, Multicenter, Phase 2 Study to Determine the Safety and Efficacy of BIND-014 (Docetaxel Nanoparticles for Injectable Suspension) as Second-line Therapy to Patients With Non-Small Cell Lung Cancer
Brief Title: A Phase 2 Study to Determine the Safety and Efficacy of BIND-014 (Docetaxel Nanoparticles for Injectable Suspension) as Second-line Therapy to Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BIND Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIND-014-005
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

ARMS (2):
- Arm A: BIND-014 every 3 weeks (Experimental)
  Interventions: Drug: BIND-014
- Arm B: BIND-014 weekly (Experimental)
  Interventions: Drug: BIND-014

INTERVENTIONS:
Drug: BIND-014

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of BIND-014 in patients with advanced non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Males or females at least 18 years of age
* Diagnosis of NSCLC with locally advanced or metastatic disease
* Previously treated with one platinum-based chemotherapy
* Disease status must be that of measurable and/or evaluable disease
* Performance status of 0 to 1 on the ECOG Scale
* Prior chemotherapy completed at least 3 weeks prior to study enrollment
* Prior radiation therapy allowed to < 25% of the bone marrow
* Patient compliance and geographic proximity that allow adequate follow-up
* Adequate organ function
* Patients with reproductive potential must use contraceptive methods
* Signed informed consent from patient

Exclusion Criteria:

* Active infection
* Pregnancy or planning to become pregnant
* Breast feeding
* Serious concomitant systemic disorders
* Second primary malignancy
* Patients who are symptomatic from brain metastasis
* Presence of detectable (by physical exam) third-space fluid collections
* More than 1 prior cytotoxic chemotherapy regimen for advanced disease
* Prior treatment with docetaxel
* History of severe hypersensitivity reaction to polysorbate 80
* Peripheral neuropathy at study entry
* Patients known to be HIV positive
* Patients known to be seropositive for hepatitis C hepatitis B
* Congenital long QT syndrome, congestive heart failure, or bradyarrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with either a complete or partial response | Patients will be followed for the duration of treatment, an expected average of 18 weeks
  To determine the efficacy of BIND-014 as measured by objective response rate (ORR) in patients with Stage III/IV Non-small cell lung cancer (NSCLC) who have failed one prior platinum containing chemotherapy regimen for advanced or metastatic disease.

SECONDARY OUTCOMES:
Number of patients who experience adverse events | Patients will be followed for the duration of treatment, an expected average of 18 weeks
  To assess the safety and tolerability of BIND-014

CONTACTS AND LOCATIONS:
Locations (17):
- United States (10):
  - Investigative Site #10, Goodyear, Arizona
  - Investigative Site #04, Los Angeles, California
  - Investigative Site #02, Fort Meyers, Florida
  - Investigative Site #08, Newnan, Georgia
  - Investigative Site #07, Zion, Illinois
  - Investigative Site #03, Columbus, Ohio
  - Investigative Site #09, Tulsa, Oklahoma
  - Investigative Site #11, Philadelphia, Pennsylvania
  - Investigative Site #05, Pittsburgh, Pennsylvania
  - Investigative Site #01, Nashville, Tennessee
- Russia (7):
  - Investigative Site #15, Chelyabinsk
  - Site #17, Krasnodar
  - Investigative Site #12, Moscow
  - Site # 18, Saint Petersburg
  - Investigative Site #14, Saint-Petersberg
  - Investigative Site #13, Saint-Petersberg
  - Investigative Site #16, Ufa

REFERENCES:
- [Background] Hrkach J, Von Hoff D, Mukkaram Ali M, Andrianova E, Auer J, Campbell T, De Witt D, Figa M, Figueiredo M, Horhota A, Low S, McDonnell K, Peeke E, Retnarajan B, Sabnis A, Schnipper E, Song JJ, Song YH, Summa J, Tompsett D, Troiano G, Van Geen Hoven T, Wright J, LoRusso P, Kantoff PW, Bander NH, Sweeney C, Farokhzad OC, Langer R, Zale S. Preclinical development and clinical translation of a PSMA-targeted docetaxel nanoparticle with a differentiated pharmacological profile. Sci Transl Med. 2012 Apr 4;4(128):128ra39. doi: 10.1126/scitranslmed.3003651. PMID 22491949